CLINICAL TRIAL: NCT03885154
Title: Valproic Acid and Dihydroergotamine as Abortive Therapy in Pediatric Migraine: An Open-Label Randomized Trial.
Brief Title: Valproic Acid and Dihydroergotamine as Abortive Therapy in Pediatric Migraine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting participants
Sponsor: Kimberly S Jones (Other)
Responsible Party: Sponsor-Investigator, Kimberly S Jones, Assistant Professor of Neurology and Pediatrics, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 44243
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Migraine in Children
Keywords: Migraine; Headache; Valproic acid; Dihydroergotamine; Pediatric
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Valproic Acid; Dihydroergotamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Valproic Acid (Active Comparator): An initial dose of Valproic Acid (VPA) will be given IV at 20mg/kg, followed by continuous infusion of 1mg/kg/hour for 24 hours. Serum levels of VPA will be checked at 4 and 24 hours, with additional timepoints possible at 8 and 12 hours based on drug levels.
  Interventions: Drug: Valproic Acid (VPA)
- Dihydroergotamine (Active Comparator): Dihydroergotamine (DHE) will be given as weight-based dosing, with no single dose >1mg and not exceeding 3mg over 24 hours.
  Interventions: Drug: Dihydroergotamine (DHE)
- Cross-Over to Dihydroergotamine (Active Comparator): An initial dose of Valproic Acid (VPA) will be given IV at 20mg/kg, followed by continuous infusion of 1mg/kg/hour for 24 hours. Serum levels of VPA will be checked at 4 and 24 hours, with additional timepoints possible at 8 and 12 hours based on drug levels. Patients who do not respond to VPA after 24 hours will be given Dihydroergotamine (DHE) for the next 24 hours. Dihydroergotamine (DHE) will be given as weight-based dosing, with no single dose >1mg and not exceeding 3mg over 24 hours.
  Interventions: Drug: Valproic Acid (VPA); Drug: Dihydroergotamine (DHE)
- Cross-Over to Valproic Acid (Active Comparator): Dihydroergotamine (DHE) will be given as weight-based dosing, with no single dose >1mg and not exceeding 3mg over 24 hours. Patients who do not respond to DHE after 24 hours will be given Valproic Acid (VPA) for the next 24 hours. An initial dose of Valproic Acid (VPA) will be given IV at 20mg/kg, followed by continuous infusion of 1mg/kg/hour for 24 hours. Serum levels of VPA will be checked at 4 and 24 hours, with additional timepoints possible at 8 and 12 hours based on drug levels.
  Interventions: Drug: Valproic Acid (VPA); Drug: Dihydroergotamine (DHE)

INTERVENTIONS:
Drug: Valproic Acid (VPA) — IV VPA load 20mg/kg, followed by continuous infusion of 1mg/kg/hr for 24 hours
  Other Names: Depakene
  Arms: Cross-Over to Dihydroergotamine; Cross-Over to Valproic Acid; Valproic Acid
Drug: Dihydroergotamine (DHE) — 0 hour: 0.50 x (wt in kg) x (0.014) =Xmg 8 hour: 0.75 x (wt in kg) x (0.014) =Xmg 24 hour: 1.00 x (wt in kg) x (0.014) =Xmg
  Arms: Cross-Over to Dihydroergotamine; Cross-Over to Valproic Acid; Dihydroergotamine

SUMMARY:
The objective of this study is to compare clinical efficacy and tolerability of valproic acid (VPA) therapy versus dihydroergotamine (DHE) as abortive therapy in pediatric migraine.

DETAILED DESCRIPTION:
The purpose of this study is to compare valproic acid (VPA) and dihydroergotamine (DHE) alone and sequentially in the treatment of pediatric migraines.

Inpatient pediatric migraine patients (based on International Classification of Headache Disorders, ICHD-II criteria) or those admitted to the University of Kentucky emergency department will receive standard of care acute headache management as per AAP/AAN guidelines. Those who fail to respond will be considered for further eligibility. Informed consent/assent will be obtained from the patients, parents or legal guardian.

Baseline labs will be collected prior to the start of the study.

1. Complete Blood Count (CBC)
2. Comprehensive Metabolic Panel (CMP)
3. Prothrombin Time/Activated Partial Thromboplastin Time/International Normalized Ratio (PT/APTT/INR)
4. Magnesium and phosphorous

Patients will initially be randomized into two groups (VPA or DHE) and treated for 24 hours. Those patients whose migraines resolve will end the study at 24 hours. Patients who are refractory to treatment will switch interventions and continue treatment for an additional 24 hours.

Intervention 1: VPA Intervention 2: DHE

Patients in Group 1 will be treated with VPA for 24 hours. They will be given an initial dose of IV VPA at 20mg/kg, followed by continuous infusion of 1mg/kg/hour for 24 hours. Serum levels of VPA will be checked at 4 and 24 hours; depending on drug levels they may also be checked at 8 and 12 hours. The target serum concentration is 100 (+/-10) ug/mL.

Patients in Group 2 will be treated with DHE for 24 hours. Dosing will be weight-based with no single dose >1mg and total 24 hour dose <3mg.

0 hour: 0.5 x (wt in kg) x (0.014) =Xmg 8 hour: 0.75 x (wt in kg) x (0.014) =Xmg 24 hour: 1.0 x (wt in kg) x (0.014) =Xmg

Patients will be assessed for migraine severity at baseline, 4, 8, 12, and 24 hours.

1. pain (using the standard 0-10 point VAS pain scale)
2. presence or absence of photophobia
3. presence or absence of phonophobia
4. presence or absence of nausea

The endpoint criterion is successful migraine resolution (improvement in VAS and resolution of photophobia, phonophobia, and nausea). Patients meeting this criterion will not continue forward in the study.

At 24 hours, those patients that are refractory to treatment will cross over to the alternate intervention, i.e. patients receiving VPA first will then get DHE, and patients receiving DHE first will then get VPA. Outcomes will be measured for the next 24 hour period as described above.

ELIGIBILITY:
Inclusion Criteria:

* acute migraine as per ICHD-II criteria
* pediatric (age 10-18)

Exclusion Criteria:

For Valproic Acid (VPA)

* Pregnancy
* Liver disease (Acute or Chronic)
* Urea Cycle Disorder
* Mitochondrial Disease

For Dihydroergotamine (DHE)

* Pregnancy
* Peripheral vascular disease, coronary heart disease
* History of cerebrovascular event
* Severe or poorly controlled hypertension
* Impaired liver or renal function
* Triptan given in last 24 hours
* Hemiplegic migraine

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valproic Acid | Dihydroergotamine | Cross-Over to Dihydroergotamine | Cross-Over to Valproic Acid
Started | 12 | 10 | 0 | 2
Completed | 12 | 10 | 0 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants where enrolled in the cross-over dihydroergotamine group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Valproic Acid | Dihydroergotamine | Cross-Over to Dihydroergotamine | Cross-Over to Valproic Acid | Total
Number analyzed (Participants) | 12 | 10 | 0 | 2 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (1.2) | 14.1 (2.0) |  | 16.0 (1.4) | 15.0 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 |  | 2 | 15
  Male | 4 | 5 |  | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0 | 0
  Asian | 0 | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0
  Black or African American | 0 | 0 |  | 0 | 0
  White | 0 | 0 |  | 0 | 0
  More than one race | 0 | 0 |  | 0 | 0
  Unknown or Not Reported | 12 | 10 |  | 2 | 24
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 |  | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Perception
Description: Change in pain perception measured by the 10-point visual analogue scale (VAS), where 0 is "no pain" and 10 is "pain as bad as it could be."
Time Frame: Baseline to 24 hours
Population: No participants were enrolled in the cross-over to dihydroergotamine arm. Participants were analyzed on a per-arm basis. Data were not collected for DHE only for the two participants who crossed over to Valproic Acid; only the combination of treatments.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Valproic Acid | Dihydroergotamine | Cross-Over to Dihydroergotamine | Cross-Over to Valproic Acid
Number analyzed (Participants) | 12 | 10 | 0 | 2
change in score on a scale | -6.2 (3.6) | -5.8 (2.9) |  | -5 (1.4)

2. Secondary Outcome: Percentage of Participants With Presence of Photophobia
Description: Presence of absence of photophobia
Time Frame: Baseline, 4, 8, 12 and 24 hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants w/photophobia
Arm/Group | Valproic Acid | Dihydroergotamine | Cross-Over to Dihydroergotamine | Cross-Over to Valproic Acid
Number analyzed (Participants) | 12 | 10 | 0 | 2
percentage of participants w/photophobia
  Baseline | 100 | 100 |  | 100
  4 hours | 58 | 42 |  | 50
  8 hours | 17 | 17 |  | 0
  12 hours | 0 | 17 |  | 0
  24 hours | 0 | 17 |  | 0

3. Secondary Outcome: Percentage of Participants With Presence of Phonophobia
Description: Presence of absence of phonophobia
Time Frame: Baseline, 4, 8, 12 and 24 hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants w/phonophobia
Arm/Group | Valproic Acid | Dihydroergotamine | Cross-Over to Dihydroergotamine | Cross-Over to Valproic Acid
Number analyzed (Participants) | 12 | 10 | 0 | 2
percentage of participants w/phonophobia
  Baseline | 100 | 92 |  | 50
  4 hours | 42 | 25 |  | 0
  8 hours | 8 | 8 |  | 0
  12 hours | 8 | 0 |  | 0
  24 hours | 0 | 0 |  | 0

4. Secondary Outcome: Percentage of Participants With Presence of Nausea
Description: Presence or absence of nausea
Time Frame: Baseline, 4, 8, 12 and 24 hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants w/nausea
Arm/Group | Valproic Acid | Dihydroergotamine | Cross-Over to Dihydroergotamine | Cross-Over to Valproic Acid
Number analyzed (Participants) | 12 | 10 | 0 | 2
percentage of participants w/nausea
  Baseline | 100 | 100 |  | 100
  4 hours | 58 | 58 |  | 0
  8 hours | 8 | 33 |  | 0
  12 hours | 8 | 33 |  | 0
  24 hours | 0 | 25 |  | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed at baseline, 4 hour, 8 hour, 12, 24 hours per intervention.
Description: No participants were enrolled in the cross-over to dihydroergotamine arm so there was no risk for all-cause mortality.
Arm/Group | Valproic Acid | Dihydroergotamine
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproic Acid (N=14) | Dihydroergotamine (N=12)
Tightness in chest (Cardiac disorders) | 0 | 2 (2) — Participant experienced chest tightness that resolved in 15 to 20 minutes
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) — Participant experienced dyspnea and anxiety

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT03885154/Prot_SAP_ICF_001.pdf